CLINICAL TRIAL: NCT06735287
Title: A Bladder-Sparing Treatment Strategies of Large-Volume Non-Muscle-Invasive Bladder Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-954
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Bladder Cancer; NMIBC
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: this study is a prospective, single-center, historical control trial, with a planned enrollment of 30 participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bladder sparing set (Experimental)
  Interventions: Procedure: bladder sparing set
- radical cystectomy set (Active Comparator)
  Interventions: Procedure: RC

INTERVENTIONS:
Procedure: bladder sparing set — after neoadjuvant chemotherapy combined with immunotherapy, maximal TURBT and a re-TURBT shall be performed then mitomycin C bladder instillation therapy will be administered
  Arms: bladder sparing set
Procedure: RC — Radical cystectomy performed immediately after three cycles of neoadjuvant therapy.
  Arms: radical cystectomy set

SUMMARY:
Bladder cancer is a common malignancy in the urinary system, ranking 11th in cancer incidence in China (3.48/100,000), with male incidence ranking 8th (5.70/100,000). It is classified as non-muscle-invasive bladder cancer (NMIBC) or muscle-invasive bladder cancer (MIBC) based on muscle involvement. About 75% of patients are initially diagnosed with NMIBC, with Ta, T1, and Tis stages comprising 70%, 20%, and 10%, respectively.

With the advancement of magnetic resonance imaging (MRI), its role in bladder cancer diagnosis and staging has expanded. Multiparametric MRI (MpMRI) enhances staging accuracy with better anatomical visualization. In 2018, Valeria et al. introduced the VI-RADS scoring system, which uses MpMRI to predict tumor stage. Retrospective studies by Wang et al. found that all tumors with a VI-RADS score of 1 were NMIBC, and 95.1% of tumors with a score of 2 were also NMIBC. A VI-RADS score of ≤2 can be used to identify NMIBC with high sensitivity.

NMIBC shows varied risks for recurrence and progression based on tumor characteristics like size, stage, grade, and multiplicity. The European Association of Urology (EAU) risk stratification system, established in 2021, classifies NMIBC into low-, intermediate-, high-, and very-high-risk groups. Transurethral resection of bladder tumor (TURBT) is the primary diagnostic and therapeutic approach for most NMIBC cases. However, residual tumors can remain after the first TURBT. For Ta and T1 tumors, 17%-72% and 33%-78% of cases show residual disease during second resection, respectively. Re-staging TURBT for T1 tumors improves prognosis. Studies show that second TURBT offers longer recurrence-free survival (47 months) compared to a single TURBT (12 months). The 5-year progression rate was 6.5% with second TURBT, compared to 23.5% with a single procedure.

Following TURBT, floating and residual tumor cells may lead to recurrence. Immediate postoperative bladder instillation of chemotherapy (e.g., pirarubicin, epirubicin, doxorubicin, mitomycin C, gemcitabine) significantly reduces recurrence in low-risk NMIBC but is less effective for intermediate- and high-risk NMIBC. For intermediate-risk NMIBC, maintenance chemotherapy is recommended, and for high-risk NMIBC, BCG immunotherapy is preferred. Both maintenance chemotherapy and BCG instillation reduce recurrence in these groups. Mitomycin C offers comparable efficacy to BCG with fewer side effects.

For patients in the very-high-risk group, immediate radical cystectomy is recommended because delayed cystectomy leads to poorer cancer-specific survival. High-risk NMIBC patients may undergo 1-3 years of BCG therapy or immediate cystectomy if necessary.

Large-volume NMIBC (≥5 cm) presents significant challenges in treatment. TURBT for large tumors often leads to difficulties in resection due to excessive bleeding, unclear vision, and increased risk of bladder wall injury. Larger tumors also increase the risk of tumor cell seeding and metastasis. Tumor size (≥3 cm) is an independent risk factor for early recurrence and progression, leading some experts to recommend immediate radical cystectomy for large-volume NMIBC.

Radical cystectomy is a high-risk procedure with complication rates of 28%-64% and mortality rates of 2.5%-2.7%. It also requires urinary diversion, which can significantly impact a patient's physical, psychological, and social well-being. Patients often face lifelong use of urinary collection devices, reducing their quality of life. Given the impact of radical cystectomy, bladder-sparing strategies have gained attention. These approaches aim to preserve the bladder while controlling tumor growth, maintaining the patient's quality of life.

Currently, no formal guidelines exist for bladder-sparing treatment of large-volume NMIBC. However, a 2022 Chinese consensus emphasizes maximal TURBT followed by adjuvant therapy to reduce recurrence and progression. Intravesical chemotherapy, particularly BCG and mitomycin C, is a key part of postoperative management. In the era of immunotherapy, PD-1/PD-L1 inhibitors are emerging as essential components of bladder-sparing strategies. Pembrolizumab, for example, has shown a 41% complete response rate in BCG-unresponsive NMIBC, leading to its FDA approval for carcinoma in situ patients who are ineligible or unwilling to undergo radical cystectomy.

Although neoadjuvant chemotherapy is not yet included in NMIBC guidelines, its success in MIBC suggests potential benefit for NMIBC. Neoadjuvant chemotherapy improves survival by 5%-10% and reduces mortality by 16%-33%. After achieving a pathological complete response (pT0), patients can avoid radical cystectomy, with a 5-year survival rate of 90%.

This study aims to explore the feasibility of bladder-sparing treatment for large-volume NMIBC, balancing quality of life with oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of large non-muscle-invasive bladder cancer: Tumor size ≥5 cm, ≤3 tumors, pre-TURBT VI-RADS score <3, or biopsy confirms non-muscle-invasive urothelial carcinoma.

Ability to tolerate neoadjuvant chemotherapy and immunotherapy: Sufficient heart, bone marrow, liver, and kidney function (according to clinical trial center normal values), no severe hematologic abnormalities or organ dysfunction (heart function 0-2, WBC ≥3.5×10⁹/L, neutrophil count ≥1.5×10⁹/L, PLT ≥75.0×10⁹/L, HGb ≥80 g/L; liver function: total bilirubin ≤1.5×ULN, AST and ALT ≤2.5×ULN; kidney function: creatinine ≤1.5×ULN, or GFR ≥60 ml/min if creatinine >1.5×ULN).

ECOG performance status: 0 or 1. No history of other malignancies. Able to receive regular mitomycin C bladder instillation therapy after TURBT. Male or female, aged ≥18 and <80 years. Voluntary participation with written informed consent, and ability to understand and comply with study requirements, including regular follow-up.

Exclusion Criteria:

* Preoperative imaging assessment with VI-RADS ≥3. Postoperative pathology showing non-urothelial carcinoma (e.g., adenocarcinoma, squamous cell carcinoma, small cell carcinoma, or mixed tumors), or urothelial carcinoma ≥T2.

Presence of lymph node and/or distant metastases. Allergy or hypersensitivity to treatment drugs, or patients with autoimmune diseases.

Any condition deemed by the investigator to potentially harm the participant or prevent them from meeting or fulfilling study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
recurrence free survival | From enrollment to 3 years post-treatment completion

SECONDARY OUTCOMES:
progress free survival | From enrollment to 3 years post-treatment completion

OTHER OUTCOMES:
overall survival | From enrollment to 3 years post-treatment completion

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China